CLINICAL TRIAL: NCT01051869
Title: A Multicentre, Randomized Trial of Simple Decompression Versus Anterior Transposition of the Ulnar Nerve for Acute, Displaced Fractures of the Distal Humerus Treated With Plate Fixation
Brief Title: Simple Decompression Versus Anterior Transposition of the Ulnar Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ulnar Nerve 06-Jan-10
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Humeral Fractures; Ulnar Nerve Compression
Keywords: distal humerus; fractures; ulnar nerve; simple decompression; anterior transposition
MeSH Terms: conditions — Humeral Fractures; Ulnar Nerve Compression Syndromes; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- simple decompression (Active Comparator)
  Interventions: Procedure: Simple decompression
- anterior subcutaneous transposition (Active Comparator)
  Interventions: Procedure: anterior subcutaneous transposition

INTERVENTIONS:
Procedure: Simple decompression — Fracture fixation will be performed through a posterior approach, as this provides excellent visualization of the distal fragments. A triceps split will be used to expose the distal humerus. A midline incision will be made from proximally to distal onto the shaft of the ulna. Equal portions of the triceps muscle will be reflected medially and laterally, with use of sharp dissection to remove the triceps insertion from the olecranon. The ulnar nerve will be identified and protected proximal and distal to the medial epicondyle. Fracture fixation will be performed after anatomic reduction using standard fixation techniques and plate fixation on both the medial and lateral column.
  In the simple ulnar nerve decompression group, no further treatment of the ulnar nerve will be undertaken.
  Arms: simple decompression
Procedure: anterior subcutaneous transposition — In the anterior transposition of the ulnar nerve group, the ulnar nerve will be placed subcutaneously anterior to the medial epicondyle free from any pressure.
  Arms: anterior subcutaneous transposition

SUMMARY:
Both simple decompression and anterior transposition of the elbow nerve (ulnar nerve) for acute displaced fractures of the elbow (distal humerus) treated with plate fixation are currently used by surgeons. We want to examine which treatment will overall give better results in regards to arm function and residual pain.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 16 to 60 years of age
* Displaced, distal humerus fracture (OTA 13A or 13C) as seen in radiographs
* Fractures ≤ 28 days post injury
* Closed fractures
* No history of previous ulnar neuropathy or elbow pathology
* Provisin of informed consent

Exclusion Criteria:

* Vascular injury
* History of previous ulnar neuropathy or elbow pathology
* Fractures more than 28 days post-injury
* Limited life expectancy due to significant medical co-morbidity or medical contraindication to surgery
* Inability to comply with rehabilitation or form completion
* Likely problems, in the judgement of the investigators, with maintaining follow-up (i.e. patients with no fixed address, patients not mentally competent to give consent, etc.)

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2010-09; Primary Completion 2018-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be signs of ulnar neuropathy, measured using two clinical staging systems to assess the degree of dysfunction of the ulnar nerve (the classification system of Gabel and Amadio13). | 1 Year

SECONDARY OUTCOMES:
Secondary outcome measurement will include a patient-oriented, limb-specific, functional measurement questionnaire (Disabilities of the Arm, Shoulder and Hand Instrument-DASH) | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Emil H Schemitsch, MD, FRCS(C), Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada